CLINICAL TRIAL: NCT04308720
Title: Circulating Tumor DNA (ctDNA) and Immunophenotyping as Potential Biomarkers in Patients Undergoing Regional Nodal Irradiation for Breast Cancer
Brief Title: Circulating Tumor DNA and Immunophenotyping as Potential Biomarkers With Regional Nodal Irradiation for Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 19-003532; NCI-2022-10695 (Registry Identifier: CTRP (Clinical Trials Reporting Program)); ROR1931 (Other: Mayo Clinic Radiation Oncology)
Record Dates: First submitted 2020-02-07; First posted 2020-03-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will assess how radiation affects the patterns of circulating tumor deoxyribonucleic acid (ctDNA) and immune cells (T cells) during radiation treatment in patients with breast cancer. By better understanding how radiation therapy affects these markers (characteristic that is measured to see how well the body responds to a treatment for a disease) in the blood, researchers may better customize treatments for patients with breast cancer in the future.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed primary or recurrent non-metastatic invasive breast cancer with plans for adjuvant post-lumpectomy or post-mastectomy radiation therapy at the Mayo Clinic and indications for regional nodal irradiation.
* Or patients undergoing curative intent irradiation for oligometastatic breast cancer (=< 3 sites of metastases) is permitted
* Willingness to provide informed consent and expresses understanding of this protocol and its requirements, risks, and discomforts
* Patients with non-metastatic breast cancer must have completed their final breast surgery including re-excision of margins for invasive cancer and ductal carcinoma in situ (DCIS) or chemotherapy within 90 days prior to registration but no sooner than 21 days prior to the initiation of radiation therapy (RT).
* Bilateral breast cancer is permitted
* Positive or close margins is allowed

Exclusion Criteria:

* Other active malignancy =< 2 years prior to registration (exceptions: non-melanotic skin cancer or carcinoma-in-situ of the cervix)
* Pregnancy or lactation
* Inability on the part of the patient to understand the informed consent to be compliant with the protocol

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women ages 18 and older with high-risk breast cancer with plan for adjuvant radiation therapy including the regional lymph nodes at Mayo Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2028-10-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Changes in the ctDNA detection | Baseline to 3 months post-treatment (treatment typically lasts 3-6 weeks)
  Assessed by the number of patients who have undetectable ctDNA post-treatment, among patients that were detectable pre-treatment.

OTHER OUTCOMES:
Explore correlation of detectable ctDNA with invasive recurrence-free survival | 3 months post-treatment (treatment typically lasts 3-6 weeks)
  Invasive recurrence is defined as the return of cancer after initial treatment, where the cancer has spread beyond the ducts or lobules into surrounding breast tissue

CONTACTS AND LOCATIONS:
Overall Officials: Robert W. Mutter, M.D., Principal Investigator — Mayo Clinic Radiation Oncology
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials